CLINICAL TRIAL: NCT06543173
Title: Primary Preventive Ventricular Tachycardia Ablation In High-Risk Patients Who Receive A Prophylactic Implantable Cardioverter Defibrillator (PRIMARY PREVENT-VT TRIAL)
Brief Title: Primary Preventive Ventricular Tachycardia Ablation In High-Risk Patients Who Receive A Prophylactic Implantable Cardioverter Defibrillator
Acronym: PREVENT-VT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Ilan Goldenberg, Ilan Goldenberg, MD, Professor of Medicine, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00009548
Record Dates: First submitted 2024-06-17; First posted 2024-08-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 fashion to undergo either prophylactic catheter-based ventricular tachycardia (VT) ablation within 3 months of primary ICD implantation or continued medical management after ICD implantation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic Catheter-based VT Ablation (Experimental): Subjects receive catheter-based ventricular tachycardia (VT) ablation within 3 months of primary ICD implantation.
  Interventions: Procedure: Prophylactic Catheter-based VT Ablation
- Continued Medical Management (No Intervention): Subjects undergo continued medical management after primary ICD implantation without prophylactic VT ablation.

INTERVENTIONS:
Procedure: Prophylactic Catheter-based VT Ablation — Prophylactic Catheter-based VT Ablation refers to a treatment strategy where participants undergo a procedure known as catheter-based ventricular tachycardia (VT) ablation shortly after receiving their primary implantable cardioverter defibrillator (ICD).
  Arms: Prophylactic Catheter-based VT Ablation

SUMMARY:
This prospective, multicenter, open-label, randomized-controlled trial compares two treatment strategies in high-risk ischemic cardiomyopathy (ICM) patients referred for primary ICD implantation. Participants will be randomized to receive either prophylactic VT ablation within three months of ICD implantation or continued medical management. The primary objective is to assess the efficacy of preventive VT ablation versus medical management in reducing VT arrhythmia burden.

DETAILED DESCRIPTION:
This study aims to assess the impact of prophylactic catheter-based ventricular tachycardia (VT) ablation compared to medical management in high-risk patients with ischemic cardiomyopathy (ICM) undergoing primary implantable cardioverter defibrillator (ICD) implantation. The primary outcome measure is the burden of VT arrhythmias (VTA), defined as the total number of VT events, one year post-ICD implantation. The hypothesis suggests that employing VT ablation with high-density electroanatomic mapping (EnsiteTM) will significantly reduce both treated and monitored VT episodes. The study will randomize 62 participants in a 1:1 ratio across 20 experienced sites in Europe.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (no upper age limit)
* Willing and able to provide informed consent
* Candidate for a primary prevention ICD/CRT-D per ESC guidelines17
* Ischemic cardiomyopathy (ICM) with left ventricular ejection fraction (LVEF) ≤ 35%
* Willing and able to receive an ICD
* Willing and able to undergo catheter-based VT ablation

One or more of the following:

* MADIT-ICD Benefit Score >75
* History of nonsustained ventricular tachycardia (NSVT)
* Multiple premature ventricular complexes (PVCs ≥10%)

Exclusion Criteria:

* Existing ICD or CRT-D
* History of sustained VT or VF
* Chronic renal failure requiring hemodialysis
* Coronary revascularization within the past 3 months
* ST-Elevation MI within the past 3 months
* Participation in concurrent clinical trials without approval from the Coordination Center (observational registries are allowed with approval)
* Currently pregnant or planning to become pregnant in the near future
* Inability or unwillingness to adhere to the study protocol
* Inability or unwillingness to provide informed consent for participation
* Life expectancy < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2030-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Total Number of VT Arrhythmia Events in High-Risk Patients with Ischemic Cardiomyopathy (ICM) After Primary ICD Implantation: Comparison of Preventive Catheter-Based VT Ablation Versus Medical Management. | One year following ICD implantation.
  Evaluating the impact of preventive catheter-based VT ablation versus medical management on the total number of VT arrhythmia events in high-risk patients with ischemic cardiomyopathy (ICM) after primary ICD implantation.

SECONDARY OUTCOMES:
Impact of Preventive VT Ablation on Healthcare Utilization, assessed using the mean rate of events per arm. | One year following ICD implantation.
  Assessing whether preventive VT ablation compared to medical management reduces healthcare resource utilization in high-risk patients with ICM after primary ICD implantation. Healthcare resource utilization will be quantified by averaging planned and unplanned in-office visits, urgent care or emergency room visits, hospitalizations, repeat ablations, or mortality per arm. Data on healthcare utilization will be collected at all follow-up visits (months 3, 6, and 9) and at the end-of-study visit. Analysis will be conducted using a t-test for comparison.

OTHER OUTCOMES:
Impact of Preventive VT Ablation on the Quality of Life Using the Kansas City Cardiomyopathy Questionnaire (KCCQ). | One year following ICD implantation.
  Assessing whether preventive VT ablation compared to medical management enhances quality of life in high-risk patients with ICM after primary ICD implantation, using the Kansas City Cardiomyopathy Questionnaire (KCCQ) to measure quality of life. Scores on the KCCQ range from 0 to 100, with higher scores indicating better quality of life. Data collection with the KCCQ will occur at the Baseline and End of Study visits. Differences in quality of life between the study groups will be analyzed using the t-test based on KCCQ responses.

REFERENCES:
- [Background] Cronin EM, Bogun FM, Maury P, Peichl P, Chen M, Namboodiri N, Aguinaga L, Leite LR, Al-Khatib SM, Anter E, Berruezo A, Callans DJ, Chung MK, Cuculich P, d'Avila A, Deal BJ, Della Bella P, Deneke T, Dickfeld TM, Hadid C, Haqqani HM, Kay GN, Latchamsetty R, Marchlinski F, Miller JM, Nogami A, Patel AR, Pathak RK, Saenz Morales LC, Santangeli P, Sapp JL Jr, Sarkozy A, Soejima K, Stevenson WG, Tedrow UB, Tzou WS, Varma N, Zeppenfeld K. 2019 HRS/EHRA/APHRS/LAHRS expert consensus statement on catheter ablation of ventricular arrhythmias: Executive summary. Heart Rhythm. 2020 Jan;17(1):e155-e205. doi: 10.1016/j.hrthm.2019.03.014. Epub 2019 May 10. PMID 31102616
- [Background] Moss AJ, Greenberg H, Case RB, Zareba W, Hall WJ, Brown MW, Daubert JP, McNitt S, Andrews ML, Elkin AD; Multicenter Automatic Defibrillator Implantation Trial-II (MADIT-II) Research Group. Long-term clinical course of patients after termination of ventricular tachyarrhythmia by an implanted defibrillator. Circulation. 2004 Dec 21;110(25):3760-5. doi: 10.1161/01.CIR.0000150390.04704.B7. Epub 2004 Dec 6. PMID 15583079
- [Background] Poole JE, Johnson GW, Hellkamp AS, Anderson J, Callans DJ, Raitt MH, Reddy RK, Marchlinski FE, Yee R, Guarnieri T, Talajic M, Wilber DJ, Fishbein DP, Packer DL, Mark DB, Lee KL, Bardy GH. Prognostic importance of defibrillator shocks in patients with heart failure. N Engl J Med. 2008 Sep 4;359(10):1009-17. doi: 10.1056/NEJMoa071098. PMID 18768944
- [Background] Schron EB, Exner DV, Yao Q, Jenkins LS, Steinberg JS, Cook JR, Kutalek SP, Friedman PL, Bubien RS, Page RL, Powell J. Quality of life in the antiarrhythmics versus implantable defibrillators trial: impact of therapy and influence of adverse symptoms and defibrillator shocks. Circulation. 2002 Feb 5;105(5):589-94. doi: 10.1161/hc0502.103330. PMID 11827924
- [Background] Noyes K, Corona E, Veazie P, Dick AW, Zhao H, Moss AJ. Examination of the effect of implantable cardioverter-defibrillators on health-related quality of life: based on results from the Multicenter Automatic Defibrillator Trial-II. Am J Cardiovasc Drugs. 2009;9(6):393-400. doi: 10.2165/11317980-000000000-00000. PMID 19929037
- [Background] Dunbar SB, Dougherty CM, Sears SF, Carroll DL, Goldstein NE, Mark DB, McDaniel G, Pressler SJ, Schron E, Wang P, Zeigler VL; American Heart Association Council on Cardiovascular Nursing, Council on Clinical Cardiology, and Council on Cardiovascular Disease in the Young. Educational and psychological interventions to improve outcomes for recipients of implantable cardioverter defibrillators and their families: a scientific statement from the American Heart Association. Circulation. 2012 Oct 23;126(17):2146-72. doi: 10.1161/CIR.0b013e31825d59fd. Epub 2012 Sep 24. PMID 23008437
- [Background] Tung R, Vaseghi M, Frankel DS, Vergara P, Di Biase L, Nagashima K, Yu R, Vangala S, Tseng CH, Choi EK, Khurshid S, Patel M, Mathuria N, Nakahara S, Tzou WS, Sauer WH, Vakil K, Tedrow U, Burkhardt JD, Tholakanahalli VN, Saliaris A, Dickfeld T, Weiss JP, Bunch TJ, Reddy M, Kanmanthareddy A, Callans DJ, Lakkireddy D, Natale A, Marchlinski F, Stevenson WG, Della Bella P, Shivkumar K. Freedom from recurrent ventricular tachycardia after catheter ablation is associated with improved survival in patients with structural heart disease: An International VT Ablation Center Collaborative Group study. Heart Rhythm. 2015 Sep;12(9):1997-2007. doi: 10.1016/j.hrthm.2015.05.036. Epub 2015 May 30. PMID 26031376
- [Background] Frankel DS, Mountantonakis SE, Robinson MR, Zado ES, Callans DJ, Marchlinski FE. Ventricular tachycardia ablation remains treatment of last resort in structural heart disease: argument for earlier intervention. J Cardiovasc Electrophysiol. 2011 Oct;22(10):1123-8. doi: 10.1111/j.1540-8167.2011.02081.x. Epub 2011 May 3. PMID 21539642
- [Background] Dinov B, Arya A, Bertagnolli L, Schirripa V, Schoene K, Sommer P, Bollmann A, Rolf S, Hindricks G. Early referral for ablation of scar-related ventricular tachycardia is associated with improved acute and long-term outcomes: results from the Heart Center of Leipzig ventricular tachycardia registry. Circ Arrhythm Electrophysiol. 2014 Dec;7(6):1144-51. doi: 10.1161/CIRCEP.114.001953. Epub 2014 Sep 27. PMID 25262159
- [Background] Reddy VY, Reynolds MR, Neuzil P, Richardson AW, Taborsky M, Jongnarangsin K, Kralovec S, Sediva L, Ruskin JN, Josephson ME. Prophylactic catheter ablation for the prevention of defibrillator therapy. N Engl J Med. 2007 Dec 27;357(26):2657-65. doi: 10.1056/NEJMoa065457. PMID 18160685
- [Background] Kuck KH, Schaumann A, Eckardt L, Willems S, Ventura R, Delacretaz E, Pitschner HF, Kautzner J, Schumacher B, Hansen PS; VTACH study group. Catheter ablation of stable ventricular tachycardia before defibrillator implantation in patients with coronary heart disease (VTACH): a multicentre randomised controlled trial. Lancet. 2010 Jan 2;375(9708):31-40. doi: 10.1016/S0140-6736(09)61755-4. PMID 20109864
- [Background] Kuck KH, Tilz RR, Deneke T, Hoffmann BA, Ventura R, Hansen PS, Zarse M, Hohnloser SH, Kautzner J, Willems S; SMS Investigators. Impact of Substrate Modification by Catheter Ablation on Implantable Cardioverter-Defibrillator Interventions in Patients With Unstable Ventricular Arrhythmias and Coronary Artery Disease: Results From the Multicenter Randomized Controlled SMS (Substrate Modification Study). Circ Arrhythm Electrophysiol. 2017 Mar;10(3):e004422. doi: 10.1161/CIRCEP.116.004422. PMID 28292751
- [Background] Willems S, Tilz RR, Steven D, Kaab S, Wegscheider K, Geller L, Meyer C, Heeger CH, Metzner A, Sinner MF, Schluter M, Nordbeck P, Eckardt L, Bogossian H, Sultan A, Wenzel B, Kuck KH; BERLIN VT Investigators. Preventive or Deferred Ablation of Ventricular Tachycardia in Patients With Ischemic Cardiomyopathy and Implantable Defibrillator (BERLIN VT): A Multicenter Randomized Trial. Circulation. 2020 Mar 31;141(13):1057-1067. doi: 10.1161/CIRCULATIONAHA.119.043400. Epub 2020 Jan 31. PMID 32000514
- [Background] Della Bella P, Baratto F, Vergara P, Bertocchi P, Santamaria M, Notarstefano P, Calo L, Orsida D, Tomasi L, Piacenti M, Sangiorgio S, Pentimalli F, Pruvot E, De Sousa J, Sacher F, Tritto M, Rebellato L, Deneke T, Romano SA, Nesti M, Gargaro A, Giacopelli D, Peretto G, Radinovic A. Does Timing of Ventricular Tachycardia Ablation Affect Prognosis in Patients With an Implantable Cardioverter Defibrillator? Results From the Multicenter Randomized PARTITA Trial. Circulation. 2022 Jun 21;145(25):1829-1838. doi: 10.1161/CIRCULATIONAHA.122.059598. Epub 2022 Apr 3. PMID 35369700
- [Background] Goldenberg I, Maury P, Huang DT, Aktas M, Sacher F, Clementy N, Mulpuru S, Friedman P, Meyer C, Tiefenbrun NL, McNitt S, Zareba W, Nof E. Hybrid VT Ablation-Subcutaneous ICD Management Strategy for Secondary Prevention of Sudden Cardiac Death: The VTabl-SICD Trial. Heart Rhythm 2023 (in press).
- [Background] Younis A, Goldberger JJ, Kutyifa V, Zareba W, Polonsky B, Klein H, Aktas MK, Huang D, Daubert J, Estes M, Cannom D, McNitt S, Stein K, Goldenberg I. Predicted benefit of an implantable cardioverter-defibrillator: the MADIT-ICD benefit score. Eur Heart J. 2021 May 1;42(17):1676-1684. doi: 10.1093/eurheartj/ehaa1057. PMID 33417692
- [Background] Zeppenfeld K, Tfelt-Hansen J, de Riva M, Winkel BG, Behr ER, Blom NA, Charron P, Corrado D, Dagres N, de Chillou C, Eckardt L, Friede T, Haugaa KH, Hocini M, Lambiase PD, Marijon E, Merino JL, Peichl P, Priori SG, Reichlin T, Schulz-Menger J, Sticherling C, Tzeis S, Verstrael A, Volterrani M; ESC Scientific Document Group. 2022 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death. Eur Heart J. 2022 Oct 21;43(40):3997-4126. doi: 10.1093/eurheartj/ehac262. No abstract available. PMID 36017572
- [Background] Arenal A, Glez-Torrecilla E, Ortiz M, Villacastin J, Fdez-Portales J, Sousa E, del Castillo S, Perez de Isla L, Jimenez J, Almendral J. Ablation of electrograms with an isolated, delayed component as treatment of unmappable monomorphic ventricular tachycardias in patients with structural heart disease. J Am Coll Cardiol. 2003 Jan 1;41(1):81-92. doi: 10.1016/s0735-1097(02)02623-2. PMID 12570949
- [Background] Jais P, Maury P, Khairy P, Sacher F, Nault I, Komatsu Y, Hocini M, Forclaz A, Jadidi AS, Weerasooryia R, Shah A, Derval N, Cochet H, Knecht S, Miyazaki S, Linton N, Rivard L, Wright M, Wilton SB, Scherr D, Pascale P, Roten L, Pederson M, Bordachar P, Laurent F, Kim SJ, Ritter P, Clementy J, Haissaguerre M. Elimination of local abnormal ventricular activities: a new end point for substrate modification in patients with scar-related ventricular tachycardia. Circulation. 2012 May 8;125(18):2184-96. doi: 10.1161/CIRCULATIONAHA.111.043216. Epub 2012 Apr 4. PMID 22492578
- [Background] Irie T, Yu R, Bradfield JS, Vaseghi M, Buch EF, Ajijola O, Macias C, Fujimura O, Mandapati R, Boyle NG, Shivkumar K, Tung R. Relationship between sinus rhythm late activation zones and critical sites for scar-related ventricular tachycardia: systematic analysis of isochronal late activation mapping. Circ Arrhythm Electrophysiol. 2015 Apr;8(2):390-9. doi: 10.1161/CIRCEP.114.002637. Epub 2015 Mar 4. PMID 25740836
- [Background] Aziz Z, Shatz D, Raiman M, Upadhyay GA, Beaser AD, Besser SA, Shatz NA, Fu Z, Jiang R, Nishimura T, Liao H, Nayak HM, Tung R. Targeted Ablation of Ventricular Tachycardia Guided by Wavefront Discontinuities During Sinus Rhythm: A New Functional Substrate Mapping Strategy. Circulation. 2019 Oct 22;140(17):1383-1397. doi: 10.1161/CIRCULATIONAHA.119.042423. Epub 2019 Sep 19. PMID 31533463
- [Background] Di Biase L, Santangeli P, Burkhardt DJ, Bai R, Mohanty P, Carbucicchio C, Dello Russo A, Casella M, Mohanty S, Pump A, Hongo R, Beheiry S, Pelargonio G, Santarelli P, Zucchetti M, Horton R, Sanchez JE, Elayi CS, Lakkireddy D, Tondo C, Natale A. Endo-epicardial homogenization of the scar versus limited substrate ablation for the treatment of electrical storms in patients with ischemic cardiomyopathy. J Am Coll Cardiol. 2012 Jul 10;60(2):132-41. doi: 10.1016/j.jacc.2012.03.044. PMID 22766340
- [Background] Soejima K, Stevenson WG, Maisel WH, Sapp JL, Epstein LM. Electrically unexcitable scar mapping based on pacing threshold for identification of the reentry circuit isthmus: feasibility for guiding ventricular tachycardia ablation. Circulation. 2002 Sep 24;106(13):1678-83. doi: 10.1161/01.cir.0000030187.39852.a7. PMID 12270862
- [Background] Tzou WS, Frankel DS, Hegeman T, Supple GE, Garcia FC, Santangeli P, Katz DF, Sauer WH, Marchlinski FE. Core isolation of critical arrhythmia elements for treatment of multiple scar-based ventricular tachycardias. Circ Arrhythm Electrophysiol. 2015 Apr;8(2):353-61. doi: 10.1161/CIRCEP.114.002310. Epub 2015 Feb 13. PMID 25681389
- [Background] Brunckhorst CB, Stevenson WG, Soejima K, Maisel WH, Delacretaz E, Friedman PL, Ben-Haim SA. Relationship of slow conduction detected by pace-mapping to ventricular tachycardia re-entry circuit sites after infarction. J Am Coll Cardiol. 2003 Mar 5;41(5):802-9. doi: 10.1016/s0735-1097(02)02932-7. PMID 12628726
- [Background] de Chillou C, Groben L, Magnin-Poull I, Andronache M, MagdiAbbas M, Zhang N, Abdelaal A, Ammar S, Sellal JM, Schwartz J, Brembilla-Perrot B, Aliot E, Marchlinski FE. Localizing the critical isthmus of postinfarct ventricular tachycardia: the value of pace-mapping during sinus rhythm. Heart Rhythm. 2014 Feb;11(2):175-81. doi: 10.1016/j.hrthm.2013.10.042. PMID 24513915
- [Background] Goldenberg I, Huang D, McNitt S, Zareba W, Aktas M, Kutyifa V. History of non-sustained ventricular tachycardia and the risk of arrhythmic events in patients with a primary prevention ICD. Heart Rhythm Scientific Sessions, 2024.
- [Background] Gopinathannair R, Cornwell WK, Dukes JW, Ellis CR, Hickey KT, Joglar JA, Pagani FD, Roukoz H, Slaughter MS, Patton KK. Device Therapy and Arrhythmia Management in Left Ventricular Assist Device Recipients: A Scientific Statement From the American Heart Association. Circulation. 2019 May 14;139(20):e967-e989. doi: 10.1161/CIR.0000000000000673. PMID 30943783
- [Background] Jamil DD, Baram A, Saqat BH. Impact of prolonged cardiopulmonary bypass and operative exposure time on the incidence of surgical site infections in patients undergoing open heart surgery: Single center case series. International Journal of Surgery Open, 2020;22:52-56.
- [Background] Brown WR, Moody DM, Challa VR, Stump DA, Hammon JW. Longer duration of cardiopulmonary bypass is associated with greater numbers of cerebral microemboli. Stroke. 2000 Mar;31(3):707-13. doi: 10.1161/01.str.31.3.707. PMID 10700508
- [Background] Mehra MR, Uriel N, Naka Y, Cleveland JC Jr, Yuzefpolskaya M, Salerno CT, Walsh MN, Milano CA, Patel CB, Hutchins SW, Ransom J, Ewald GA, Itoh A, Raval NY, Silvestry SC, Cogswell R, John R, Bhimaraj A, Bruckner BA, Lowes BD, Um JY, Jeevanandam V, Sayer G, Mangi AA, Molina EJ, Sheikh F, Aaronson K, Pagani FD, Cotts WG, Tatooles AJ, Babu A, Chomsky D, Katz JN, Tessmann PB, Dean D, Krishnamoorthy A, Chuang J, Topuria I, Sood P, Goldstein DJ; MOMENTUM 3 Investigators. A Fully Magnetically Levitated Left Ventricular Assist Device - Final Report. N Engl J Med. 2019 Apr 25;380(17):1618-1627. doi: 10.1056/NEJMoa1900486. Epub 2019 Mar 17. PMID 30883052